CLINICAL TRIAL: NCT01923441
Title: Evaluation of the Effectiveness and Clinical Utility of Brain Network Activation (BNA™) Technology in the Management of Sport Related Concussion in Youth and Adolescents Athletes.
Status: Completed | Type: Observational
Sponsor: ElMindA Ltd (Industry)
Collaborators: Athletico Physical Therapy (Other)
Responsible Party: Sponsor
Other Study IDs: ELM-21
Record Dates: First submitted 2013-08-13; First posted 2013-08-15 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2013-08

CONDITIONS: Minor Traumatic Brain Injury (TBI)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Highschool athletes
- midschool athletes

SUMMARY:
Currently, there is no direct, reliable, bed-side, and non-invasive method for assessing changes in brain activity associated with concussion. Event Related Potentials (ERPs), which are temporal reflections of the neural mass electrical activity of cells in specific regions of the brain that occur in response to stimuli, may offer such a method, as they provide both a noninvasive and portable measure of brain function. The ERPs provide excellent temporal information, but spatial resolution for ERPs has traditionally been limited. However, by using high-density electroencephalograph (EEG) recording spatial resolution for ERPs is improved significantly. The paradigm for the current study will combine neurophysiological knowledge with mathematical signal processing and pattern recognition methods (BNA™) to temporally and spatially map brain function, connectivity and synchronization.

The proposed study will provide additional evidence for the utility and contribution of the BNA™ test (reflecting temporal and spatial changes in brain activity as well as brain functional connectivity associated with concussion) in concussion management.

ELIGIBILITY:
Inclusion Criteria:

* Athletes Ages 10-19, both genders, enrolled in Nazareth Academy , Deerfield High School or the Deerfield young warriors youth Football program .

Exclusion Criteria:

* Self-reported history of central nervous system injury or disease (examples will include, but will not be limited to, moderate or severe traumatic brain injury (TBI with a Glasgow Coma Scale < 13), epilepsy, seizures, brain surgery, or any positive neuroimaging results)
* Active head lice infection, open scalp wound
* deafness, and/or blindness
* Sustained a concussion within six months
* Residual symptoms or deficits related to a previous concussion
* Long and thick hair that prevents the proper administration of an EEG cap.

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Up to 300 athletes from Nazareth Academy, Deerfield High School and the Deerfield young warriors program athletes, from both genders, aged 10-19 years
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2013-08; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Changes in BNA™ measures during the sport season in both concussed and non concussed athletes compared to pre season BNA™ baseline measures. | 1 year
Correlation of the BNA measures during the sport season in both concussed and non concussed athletes to the clinical diagnosis, symptom scores and the ImPACT test results. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mike Palm, MS,MBA, Principal Investigator — Athletico Physical Therapy
Locations (1):
- Athletico N. LaGrange Rd, La Grange Park, Illinois, United States